CLINICAL TRIAL: NCT03645876
Title: SHR-1210，a Novel Anti-pd-1 Antibody, in Combination With BP102,a Biosimilar of Bevacizumab, and XELOX, (Oxaliplatin Plus Capecitabine) in Patient With Metastatic Colorectal Cancer: a Single-arm, Open Label, Multi-center, Phase II Study
Brief Title: SHR-1210 in Combination With BP102 and XELOX in Patient With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to company decision
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-210
Record Dates: First submitted 2018-08-20; First posted 2018-08-24 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: SHR-1210; BP102; Phase II
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210+BP102+XELOX (Experimental): Participants receive SHR-1210 200mg,BP102 7.5mg/kg and oxaliplatin 130mg/m2 in day 1 intravenously every 3week, capecitabine by oral bid in day1-14 every 3 week until disease progression or unacceptable toxicity
  Interventions: Drug: SHR-1210; Drug: BP102; Drug: oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: SHR-1210 — 200mg
Drug: BP102 — 7.5mg/kg
Drug: oxaliplatin — 130mg/m2
Drug: capecitabine — 1000mg/m2

SUMMARY:
This is an open label, single-arm, multi-center, phase II study of SHR-1210 in metastatic colorectal cancer patients with the recurrent lesion(s) post-surgery or the untreated mCRC.

SHR-1210 is a humanized monoclonal antibody against Programmed death 1(PD-1).BP102 is a humanized recombinant monoclonal IgG1 antibody.

The primary objective of this study is to investigate the safety and efficacy of the subjects who given the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75 years old;
2. Histologically confirmed colorectal cancer with a metastatic / recurrent lesion that cannot be cured by surgery.
3. At least one measurable lesion have been the confirmatory detection respect to RECIST 1.1
4. No prior first-line systemic anti-tumor therapy for mCRC (including systemic chemotherapy, molecular targeted therapy, biotherapy, immunotherapy, radiotherapy, local therapy and other study treatment) have been identified
5. At least 6 months have elapsed if considering the interval from the time of firstly documented metastasis to the post-operational adjuvant chemotherapy termination
6. Can provide either a newly obtained or archival tumor tissue sample.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
8. Life expectancy ≥ 3 months
9. Subjects must have normal organ and marrow function as defined below:

   1. Absolute neutrophil count (ANC) ≥1,500 /mm3（1.5×109 /L）
   2. Platelets ≥90,000 / mm3（90×109 /L）
   3. Hemoglobin ≥10 g/dL, within the 2 weeks prior to the screening no need for the transfusion
   4. Serum albumin ≥2.8 g/dL
   5. Total bilirubin≤ 1.5 X ULN, AST (SGOT), ALT (SGPT) ≤ 2.5 X ULN (AST/ALT ≤ 5 X ULN if liver metastatic);
   6. Creatinine clearance ≥ 50 mL/min according to Cockcroft-Gault formula
10. For females of child bearing potential, a negative urine or serum pregnancy test result within 72h before study treatment. Participants of reproductive potential must be willing to use adequate contraception for the course of the study until 3 months after the last dose of any of the drugs in the study.
11. The subjects are accredited with good compliance, signed the informed consent, and capable to cooperate, completing the relevant examination and follow-ups.

Exclusion Criteria:

1. Prior first-line systemic anti-tumor therapy for mCRC (including systemic chemotherapy, molecular targeted therapy, immunotherapy, biotherapy, and other treatment).
2. The metastatic/recurrent lesion is subject to be cured by surgical intervention.
3. Major operation or open biopsy or major trauma within 4 weeks prior to first dose.
4. Known Cerebral and/or leptomeningeal metastasis.
5. Bleeding predisposition, high bleeding risk or coagulant disorder, thrombotic event(s) occurrence ≤6 months and/or hemoptysis ≤3 months (≥ 1/2 teaspoons fresh blood each) prior to the screening; use of full dose oral or parenteral anticoagulant or thrombolytic medication (allowing preventative anticoagulation); use of aspirin (> 325 mg/day) or other platelet-inhibition non-steroidal anti-inflammatory drugs within 10 days since the screening; CT/MRI imaging evidence, testimony of the main arteries/veins (such as pulmonary artery or superior vena cava) being infringed, encroached
6. Subjects with uncontrolled hypertension and with a medical history of hypertensive crisis or hypertensive encephalopathy; serious cardiovascular and cerebrovascular diseases, including cerebrovascular accident (CVA) ≤6 months before the screening, transient ischemic attack (TIA), myocardial infarction and significant vascular disease (including but not limited to aortic aneurysms with need for surgical repair or recent evidence of arterial thrombosis), unstable angina, heart failure and serious arrhythmias that are uncontrolled by drugs (New York Heart Association Class ≥2).
7. Subjects with non-healing wounds, active peptic ulcer or fracture and active infection; tracheal esophageal fistula, gastrointestinal perforation or gastrointestinal fistula and abdominal abscess in the 6 months prior to the screening.
8. Subjects with any active autoimmune disease or history of autoimmune disease
9. Active infection or an unexplained fever > 38.5°C before two weeks of randomization (subjects with tumor fever may be enrolled at the discretion of the investigator);
10. History of Interstitial Pneumonia or received Corticosteroids for non-infectious pneumonitis.
11. Known Human Immunodeficiency Virus (HIV) infection、active Hepatitis B or Hepatitis C.
12. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR-1210 or BP102 formulation, allergy, hypersensitivity, or contraindication to oxaliplatin, or Capecitabine
13. Currently participating or has participated in a study within 4 weeks of the first dose of study medication.
14. Has a known additional malignancy within the last 5 years before study treatment with the exception of curatively treated basal cell and squamous cell carcinoma of the skin and/or curatively resected in-situ cervical and/or breast cancers
15. Received a live vaccine within 4 weeks of the first dose of study medication
16. Pregnancy or breast feeding.
17. According to the investigator, other conditions that may lead to stop the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Safety of the combination therapy: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 24 months
  From sign icf to the end of follow-up
Objective response rate | 24 months
  From sign icf to occurrence of objective response (complete regression (CR) and partial regression (PR) need to be confirmed 28 days after the occurrence)

SECONDARY OUTCOMES:
DOR | 24 months
  Duration of response ,DOR
DCR | 24 months
  Disease Control Rate，DCR
PFS | 24 months
  Progression free survival,PFS
9month PFS rate | 9 months
  Month 9 PFS rate,PFS9m
12month and 24 month OS rate | 24 months
  Overall survival rate: the time from the date of icf to the date of documented clinical or radiological progression or death due to any cause within 12 and 24 months after first visit

OTHER OUTCOMES:
Biomarkers and ADA | 24 months
  PD-L1、MSI、TMB expression and ADA

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No